CLINICAL TRIAL: NCT00809991
Title: Hypofractionated Adaptive Image-Guided Radiation Therapy for Localized Adenocarcinoma of the Prostate
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0859; NA_00019393 (Other: JHM IRB)
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hypofractionated radiation therapy in prostate adenocarcinoma (Experimental): Participants with histologically confirmed, locally confined adenocarcinoma of the prostate receive 3.6 Gy per day to a total dose of 57.6 Gy (16 fractions).
  Interventions: Radiation: hypofractionation

INTERVENTIONS:
Radiation: hypofractionation — 3.6 Gy per day to a total dose of 57.6 Gy (16 fractions). T

SUMMARY:
This will be a Phase II study evaluating the effectiveness and toxicity of a specific radiation therapy regimen. This choice of daily dose is based on the prior published experience showing safety and efficacy of hypofractionated regimens. The total dose is calculated to be effective for late effects which has been shown to be effective and safe in a large prospective Phase II study. If the hypothesis for the prostate is is true, then this regimen should be at least as effective or more effective for tumor control than the current conventional therapy.

DETAILED DESCRIPTION:
Radiation therapy is an effective and frequently utilized modality for the treatment of clinically localized prostate cancer. Traditionally, external beam radiation has been delivered in a fractionated manner using daily doses of 1.8-2.0 Gy. This daily dose was derived from early animal experiments and clinical experience, supported by mathematical models of normal tissue and tumor response to fraction size. The most widely used of these models is the linear-quadratic formula, which predicts responses to different fraction sizes based on the alpha/beta ratio of any given tissue.

One of the main motivations for delivering a treatment at low dose rate or with many fractions is that late-responding normal tissue are generally more sensitive than early-responding tissues (i.e. tumor) to increases in fraction size. So increasing the number of fractions generally spares late-responding tissues more than the tumor. This can be quantified in terms of the alpha/beta ratio:

* Small alpha/beta ratio (2-4 Gy), typical of late sequelae, means high sensitivity to fractionation changes.
* Large alpha/beta ratio (>8 Gy), typical of tumor control, means low sensitivity to fractionation changes.

It is generally assumed that the mechanistic basis for the different fractionation response of tumors and late-responding normal tissues relates to the larger proportion of cycling cells in tumors. But prostate tumors contain unusually small fractions of cycling cells. Brenner and Hall as well as Duchesne and Peters have reasoned that prostate tumors might not respond to changes in fractionation in the same way as other cancers; both papers hypothesize that prostate tumors might respond to changes in fractionation or dose rate more like a late-responding normal tissue. , In mathematical terms, the suggestion is that the alpha/beta ratio for prostate cancer might be low, comparable to that for late-responding tissues or even lower. Previous estimates of alpha/beta ratios of normal tissue and tumor tissue have generally been 3 and 10, respectively. Recent evidence has estimated the alpha/beta ratio of prostate cancer to be as low as 1.5. If these hypotheses are true, then the optimal therapeutic ratio for prostate cancer would be achieved using daily doses higher than 2 Gy.

Several preliminary clinical reports have found reasonable PSA control rates and no increase in late toxicity using doses of 2.5 to 3 Gy. Kupelian from the Mayo Clinic found PSA-free survival rates of 97%, 88%, and 70% in low-, intermediate-, and high-risk patients, respectively. The dose regimen used was 70 Gy in 2.5 Gy daily fractions. Both acute and late toxicity were not higher than seen with typical dose regimens. A group from Christie Hospital reported 82%, 56%, and 39% 5-year biochemical disease free survival rates (low, intermediate, and high risk, respectively) in patients treated with 50 Gy in 16 fractions (3.125 Gy per fraction), with acceptable bowel and bladder toxicity.

These results, although promising, require further validation. If the hypothesis that prostate cancer alpha/beta ratio is lower than normal tissue is correct, then the optimal fractional dose is likely to be even higher than the doses tested thus far, but if incorrect, the result may be increased normal tissue toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, locally confined adenocarcinoma of the prostate
* Clinical stages T1a to T2b PSA of less than 10 ng per ml
* Gleason score of less than 3+4=7
* The patient has decided to undergo external beam radiation as treatment choice for his prostate cancer
* Signed study-specific consent form prior to registration

Exclusion Criteria:

* Stage T3 to 4 disease
* Gleason 4+3=7 or higher score
* PSA greater than 10 ng per ml
* Clinical or Pathological Lymph node involvement N1
* Evidence of distant metastases M1
* Radical surgery for carcinoma of the prostate
* Previous Chemotherapy or pelvic radiation therapy
* Previous or concurrent cancers other than basal or squamous cell skin cancers or superficial bladder cancer unless disease free for at least 5 years
* History of inflammatory bowel disease
* Major medical or psychiatric illness which, in the investigator's opinion, would prevent completion of treatment and would interfere with follow up

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2008-12-22 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Assess the incidence of grade 2 or greater GU and GI toxicity and self-reported quality of life data with image-guided radiation therapy in doses of 3.6 Gy per day to a total dose of 57.6Gy (16 fractions). | 7 years

SECONDARY OUTCOMES:
Assess biochemical and clinical control rates associated with the hypofractionated dose regimen for both low-risk and intermediate-risk groups. Assessment will be performed at median 4 years and again at median 7 years' follow-up. | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Danny Song, MD, Principal Investigator — The Johns Hopkins University School of Medcine
Locations (1):
- The Johns Hopkins University School of Medicne, Baltimore, Maryland, United States